CLINICAL TRIAL: NCT03044223
Title: Phenotypical Und Functional Characterization of Macrophages in Critically Ill Patients With Pseudomonas Aeruginosa Induced Sepsis
Brief Title: Monocyte Profiles in Critically Ill Patients With Pseudomonas Aeruginosa Sepsis
Acronym: MIPSA
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, University of Ulm
Other Study IDs: PSA_Sepsis_M_1_2
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pseudomonas Infections; Pseudomonas Septicemia; Pseudomonas; Pneumonia; Pseudomonal Bacteraemia; Pseudomonas Urinary Tract Infection; Pseudomonas Gastrointestinal Tract Infection; Sepsis; Sepsis, Severe; Critically Ill
Keywords: pseudomonas aeruginosa; critically ill patient; sepsis; monocyte; macrophage; cytokine; severity of disease
MeSH Terms: conditions — Pseudomonas Infections; Pneumonia; Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study focuses on patients with Pseudomonas aeruginosa (PSA) sepsis. The aim of the present study is to find out whether the M1 (pro-inflammatory) or M2 (anti-inflammatory) phenotype predominates in blood monocytes in critically ill patients with PSA-sepsis, and whether the severity of sepsis and outcome is associated with distinct monocyte phenotype and function.

DETAILED DESCRIPTION:
During bacterial related sepsis, one of the key playing cells are macrophages, monocytes and T-lymphocytes (Hotchkiss et al., 2003). Macrophages and monocytes are supposed to be essential for the septic reaction to Gram-negative bacteria (Hotchkiss et al. 2003). Generally, there are two dominant types of macrophages: the pro-inflammatory M1 macrophage and the anti-inflammatory M2 macrophage (Mantovani et al., 2006). Similar to this macrophage characteristics, monocytes can also be categorized into pro-or anti-inflammatory. These macrophage/monocyte phenotypes can be differentiated in vitro from freshly isolated human blood monocytes using either GM-CSF giving raise to M1 macrophage/monocyte or M-CSF resulting in M2 macrophage/monocyte (Mantovani et al., 2006; Neu et al., 2013). Brunialti et al. (2012) have already demonstrated that the population of antiinflammatory M2 monocytes in septic patients is bigger than the pro-inflammatory M1 population. However, the authors did not further analyze the underlying mechanisms of M2 polarization nor did they identify the sepsis-causing pathogens.

In the present study, monocytes and macrophages of patients with Pseudomonas aeruginosa (PSA) sepsis are characterized by their surface marker expression profile via flow cytometry and cytokine pattern by ELISA in vivo and after ex-vivo LPS stimulation. In addition, an ex-vivo model system for PSA induced sepsis is validated. Blood of critically ill patients in the ICU infected with PSA is sampled to isolate peripheral blood mononuclear cells (PBMCs). Blood monocytes are analyzed for surface marker expression to determine the relative proportions of M1 and M2 monocytes in these patients and in healthy controls by flow cytometry

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* critically ill patients with sepsis
* microbiologically proven infection with Pseudomonas aeruginosa

Exclusion Criteria:

* life expectancy < 24 hours
* participation in other studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis with microbiologically proven infection with Pseudomonas aeruginosa
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Monocyte surface marker expression in critically ill patients with Pseudomonas aeruginosa sepsis | two years
  Monocyte type 1, type 2 surface marker expression

SECONDARY OUTCOMES:
Cytokine concentrations in serum and production after ex-vivo stimulation of isolated monocytes of critically ill patients with Pseudomonas aeruginosa sepsis with LPS | four years
  IL-8 and IFN-gamma

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, MBA, Principal Investigator — University Ulm, University Hospital Ulm; Anne Sedlag, Biochemist, Principal Investigator — University Ulm, Institute of Microbiology and Biotechnology
Locations (1):
- Clinic of Anesthesiology, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunialti MK, Santos MC, Rigato O, Machado FR, Silva E, Salomao R. Increased percentages of T helper cells producing IL-17 and monocytes expressing markers of alternative activation in patients with sepsis. PLoS One. 2012;7(5):e37393. doi: 10.1371/journal.pone.0037393. Epub 2012 May 31. PMID 22693573
- [Background] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Background] Mantovani A, Sica A, Locati M. New vistas on macrophage differentiation and activation. Eur J Immunol. 2007 Jan;37(1):14-6. doi: 10.1002/eji.200636910. PMID 17183610
- [Result] Neu C, Sedlag A, Bayer C, Forster S, Crauwels P, Niess JH, van Zandbergen G, Frascaroli G, Riedel CU. CD14-dependent monocyte isolation enhances phagocytosis of listeria monocytogenes by proinflammatory, GM-CSF-derived macrophages. PLoS One. 2013 Jun 11;8(6):e66898. doi: 10.1371/journal.pone.0066898. Print 2013. PMID 23776701